CLINICAL TRIAL: NCT03834740
Title: A Phase 0/I Study of Ribociclib (LEE011) in Combination With Everolimus in Preoperative Rb-Intact Recurrent High-Grade Glioma Patients Scheduled for Resection to Evaluate Central Nervous System (CNS) Penetration
Brief Title: A Phase 0/I Study of Ribociclib (LEE011) in Combination With Everolimus in Preoperative Recurrent High-Grade Glioma Patients Scheduled for Resection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Ivy Brain Tumor Center (Other); Barrow Neurological Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-500-311-70-38
Record Dates: First submitted 2019-01-30; First posted 2019-02-08 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma Multiforme; Glioma of Brain
Keywords: recurrent GBM; brain tumor; GBM; glioma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — ribociclib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: last dose 1 to 3 hours prior to resection (Experimental): Three to fourteen patients will receive ribociclib and everolimus orally-administered in 5 daily doses with the last dose being administered at one of 3 intervals before brain tumor resection:
  • Cohort 1: last ribociclib+everolimus dose 1 to 3 hours prior to craniotomy for tumor resection
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Cohort 2: last dose 7 to 9 hours prior to resection (Experimental): Three to fourteen patients will receive ribociclib and everolimus orally-administered in 5 daily doses with the last dose being administered at one of 3 intervals before brain tumor resection:
  • Cohort 2: last ribociclib+everolimus dose 7 to 9 hours prior to craniotomy for tumor resection
  Interventions: Drug: Ribociclib; Drug: Everolimus
- Cohort 3: last dose 23 to 25 hours prior to resection (Experimental): Three to fourteen patients will receive ribociclib and everolimus orally-administered in 5 daily doses with the last dose being administered at one of 3 intervals before brain tumor resection:
  • Cohort 3: last ribociclib+everolimus dose 23 to 25 hours prior to craniotomy for tumor resection
  Interventions: Drug: Ribociclib; Drug: Everolimus

INTERVENTIONS:
Drug: Ribociclib — Ribociclib administered orally in 5 daily doses prior to resection
Drug: Everolimus — Everolimus administered orally in 5 daily doses prior to resection

SUMMARY:
In the proposed trial, patients will be administered ribociclib+everolimus prior to surgical resection of their tumor. Recurrent GBM patients will be randomized into one of the three time-interval cohorts for the first two dose levels.

In the lead-in dose escalation study, the first six subjects (lead-in) will receive ribociclib 400 mg and everolimus 2.5 mg orally-administered in 5 daily doses with the last dose. If one or less patient experiences DLT among the 6 patients, this regimen with ribociclib 400 mg and everolimus 2.5mg will be considered safe and we will continue with the dose escalation phase of the study up to Level 3.

Four dose escalation levels:

Level 0: ribociclib 400mg and everolimus 2.5

Level 1: ribociclib 600mg and everolimus 2.5mg

Level 2: ribociclib 600mg and everolimus 5mg

Level 3: ribociclib 600mg and everolimus 10mg

ELIGIBILITY:
Inclusion Criteria:

1. Prior resection of histologically-diagnosed WHO Grade III or IV glioma. A. Glioma patients who have progressed on or following standard (Stupp regimen) therapy, which included maximal surgical resection, temozolomide, and fractionated radiotherapy.
2. Recurrence must be confirmed by diagnostic biopsy with local pathology review or contrast-enhanced MRI.
3. Subjects must have measurable disease preoperatively, defined as at least 1 contrast-enhancing lesion, with 2 perpendicular measurements of at least 1 cm, as per RANO criteria.
4. For gliomas, archival tissue must demonstrate: (a) RB positivity (≥20%) on immunohistochemistry OR no RB mutations on next-generation sequencing (NGS), (b) Chromosomal loss of CDKN2A/B/C OR CDK4/6 or CCND1/2 amplification on array CGH, (c) mTOR+: PTEN loss OR PIK3C2B or AKT3 amplification on aCGH OR mutations for PIK3CA or PIK3R1, or mTOR or PTEN mutations using rhAMP analysis or pS6 positivity on immunohistochemistry (≥10% for pS6). If mutations within the mTOR/PI3K pathways cannot be accurately detected due to poor tissue quality the enrollment criteria will be determined using RB and pS6 positivity.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Appendix 1)
6. Patients ≥ 18 years of age
7. Ability to understand and the willingness to sign a written informed consent document. (personally or by the legally authorized representative, if applicable).
8. Patient has voluntarily agreed to participate by giving written informed consent.(personally or by the legally authorized representative, if applicable).

   (Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.)
9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
10. Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or patient has had a hysterectomy.
11. Patient has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

    The following laboratory criteria have been met:
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (recommended)
    * Hemoglobin (Hgb) ≥ 9.0 g/dL
    * Platelets ≥ 100 x 109/L
    * Potassium, total calcium (corrected for serum albumin), magnesium, sodium, and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication.
    * INR ≤1.5 (unless the patient is receiving anticoagulants and the INR is within the therapeutic range of intended use for that anticoagulant within 7 days prior to the first dose of study drug)
    * Serum creatinine < 1.5 mg/dL
    * Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min.
    * In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN.
    * Serum total bilirubin <ULN, or < 3.0 x ULN in patients with well-documented Gilbert's syndrome.
    * Serum cholesterol < 300 mg/dL or < 7.75 mmol/L AND triclycerides < 2.5 x ULN (NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.)
12. QTcF interval at screening < 450 msec [using Fridericia's correction (formula = QT/(RR)0.33)]
13. Resting heart rate 50-90 bpm (may be repeated up to 2x)
14. Must be able to swallow ribociclib and everolimus capsules/tablets

Exclusion Criteria:

Patients eligible must not meet any of the following criteria:

1. Archival tissue is not available for research use or there is not a sufficient quantity available to confirm eligibility.
2. Archival tumor is not Rb-positive status and mTOR-positive status
3. Patient has not received prior radiotherapy
4. Co-morbid condition(s) that, at the opinion of the investigator, prevent safe surgical treatment
5. Active infection or fever > 38.5°C
6. Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA)
7. Known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air)
8. Active, bleeding diathesis
9. Patients with known hypersensitivity to any of the excipients of ribociclib or mTOR inhibitors (sirolimus or everolimus), including peanut, soy and lactose
10. Patients with a clinically significant hypersensitivity to everolimus or to other rapamycin derivatives.
11. Prior therapy with ribociclib or any CDK4/6 inhibitor (e.g. palbociclib, abemaciclib), or with everolimus
12. Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated
13. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer
14. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
15. Patient has a known history of HIV infection (seropositivity; testing not mandatory)
16. Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines
17. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
18. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy as indicated by the medical history. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
19. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    * Documented cardiomyopathy
    * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
    * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
    * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
    * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
    * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening (may be repeated up to 2x).
20. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Appendix 2 for details):

    * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, pomegranates or pomegranate juice and Seville oranges
    * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
    * Herbal preparations/medications, dietary supplements known as strong inhibitors or inducers of CYP3A4 or those with a known risk of QT prolongation. (Does not include Ca, Mg, Vit D or KCl supplements)
    * Known strong inhibitors or inducers of P-gp
21. Patients taking ACE inhibitors
22. Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed
23. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
24. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
25. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade ≤2 (Exception to this criterion: patients with any grade of alopecia and amenorrhea are allowed to enter the study)
26. Patient with a Child-Pugh score B or C
27. Patient has a history of non-compliance to medical regimen or inability to grant consent
28. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.]
29. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unwilling to use highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
    * In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment
    * Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
30. Sexually active males unwilling to use a condom during intercourse while taking drug and for 21 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Deputy Director of the Ivy Brain Tumor Center
Locations (3):
- United States (3):
  - Chandler Regional Medical Center, Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson KC, Tien AC, Jiang J, McNamara J, Chang YW, Montgomery C, DeSantis A, Elena-Sanchez L, Fujita Y, Kim S, Spitzer A, Gabriel P, Flynn WF, Courtois ET, Hong A, Harmon J, Umemura Y, Tovmasyan A, Li J, Mehta S, Verhaak RGW, Sanai N. Single nucleus transcriptomics, pharmacokinetics, and pharmacodynamics of CDK4/6 and mTOR inhibition in a phase 0/1 trial of recurrent high-grade glioma. Neuro Oncol. 2025 Nov 8:noaf257. doi: 10.1093/neuonc/noaf257. Online ahead of print. PMID 41206763
- [Derived] Johnson KC, Tien AC, Jiang J, McNamara J, Chang YW, Montgomery C, DeSantis A, Elena-Sanchez L, Fujita Y, Kim S, Spitzer A, Gabriel P, Flynn WF, Courtois ET, Hong A, Harmon J, Umemura Y, Tovmasyan A, Li J, Mehta S, Verhaak R, Sanai N. Single nucleus transcriptomics, pharmacokinetics, and pharmacodynamics of combined CDK4/6 and mTOR inhibition in a phase 0/1 trial of recurrent high-grade glioma. medRxiv [Preprint]. 2024 Jun 7:2024.06.07.24308439. doi: 10.1101/2024.06.07.24308439. PMID 38883740

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 enrolled participants were assigned to 1 of 7 different dose escalation levels of ribociclib plus everolimus. For all levels, ribo doses were administered orally QD for five days. For levels 0-3, eve doses were administered orally QD for five days. For levels 4-6, a single dose of eve was administered once on day 5. Participants were also assigned to 1 of 3 time interval cohorts, each with a different timing for the administration of the final dose combination before brain tumor resection.
Groups:
- Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy: The final of five ribociclib+everolimus doses administered orally 1 to 3 hours prior to craniotomy for tumor resection
- Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy: The final of five ribociclib+everolimus doses administered orally 7 to 9 hours prior to craniotomy for tumor resection
- Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy: The final of five ribociclib+everolimus doses administered orally 23 to 25 hours prior to craniotomy for tumor resection
Period: Ribo 400mg+Eve 2.5mg QD
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Ribo 600mg+Eve 2.5mg QD
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 1 | 2 | 0
Completed | 1 | 2 | 0
Not Completed | 0 | 0 | 0
Period: Ribo 600mg+Eve 5mg QD
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Ribo 600mg+Eve 10mg QD
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 0 | 4 | 0
Completed | 0 | 4 | 0
Not Completed | 0 | 0 | 0
Period: Ribo 600mg QD+Eve 50mg Once
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 0 | 4 | 0
Completed | 0 | 4 | 0
Not Completed | 0 | 0 | 0
Period: Ribo 600mg QD+Eve 60mg Once
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Ribo 600mg QD+Eve 70mg Once
Arm/Group | Time Cohort 1: Final Dose 1 to 3 Hours Prior to Craniotomy | Time Cohort 2: Final Dose 7 to 9 Hours Prior to Craniotomy | Time Cohort 3: Final Dose 23 to 25 Hours Prior to Craniotomy
Started | 0 | 4 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 27 enrolled participants were included in safety and tolerability analysis
Groups:
- Dose Level 0: Ribo 400mg+Eve 2.5mg QD: Dose Level 0: Ribo 400mg+Eve 2.5mg QD and all 3 Time Cohorts were combined
- Dose Level 1: Ribo 600mg+Eve 2.5mg QD: Dose Level 1: Ribo 600mg+Eve 2.5mg QD of participants in both Time Cohorts 1 and 2 as only 1 participant in Time Cohort 1 at this dose level
- Dose Level 2: Ribo 600mg+Eve 5mg QD: Dose Level 2: Ribo 600mg+Eve 5mg QD of participants in Time Cohort 2
- Dose Level 3: Ribo 600mg+Eve 10mg QD: Dose Level 3: Ribo 600mg+Eve 10mg QD of participants in Time Cohort 2
- Dose Level 4: Ribo 600mg QD+Eve 50mg Once: Dose Level 4: Ribo 600mg QD+Eve 50mg Once of participants in Time Cohort 2
- Dose Level 5: Ribo 600mg QD+Eve 60mg Once: Dose Level 5: Ribo 600mg QD+Eve 60mg Once of participants in Time Cohort 2
- Dose Level 6: Ribo 600mg QD+Eve 70mg Once: Dose Level 6: Ribo 600mg QD+Eve 70mg Once of participants in Time Cohort 2
- Total: Total of all reporting groups
Arm/Group | Dose Level 0: Ribo 400mg+Eve 2.5mg QD | Dose Level 1: Ribo 600mg+Eve 2.5mg QD | Dose Level 2: Ribo 600mg+Eve 5mg QD | Dose Level 3: Ribo 600mg+Eve 10mg QD | Dose Level 4: Ribo 600mg QD+Eve 50mg Once | Dose Level 5: Ribo 600mg QD+Eve 60mg Once | Dose Level 6: Ribo 600mg QD+Eve 70mg Once | Total
Number analyzed (Participants) | 6 | 3 | 3 | 4 | 4 | 3 | 4 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 1 | 4 | 1 | 3 | 4 | 20
  >=65 years | 1 | 1 | 2 | 0 | 3 | 0 | 0 | 7
Age, Continuous [Median (Full Range); unit: Years] | 54 [34 to 70] | 58 [52 to 70] | 65 [58 to 65] | 54.5 [45 to 58] | 68 [61 to 72] | 61 [46 to 63] | 49 [35 to 58] | 58 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 1 | 2 | 2 | 8
  Male | 4 | 2 | 3 | 4 | 3 | 1 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 6 | 2 | 3 | 4 | 4 | 2 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 2 | 3 | 4 | 4 | 3 | 4 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Highest dose of each drug that did not cause a DLT in >17% of participants
Time Frame: From the date of the first dose given until the second documented DLT, assessed up to 24 months
Population: Enrolled participants
Measure: Number; unit: milligrams
Groups:
- All Participants: All participants enrolled in the clinical trial.
Arm/Group | All Participants
Number analyzed (Participants) | 24
milligrams
  Ribociclib, once daily | 600
  Everolimus, once weekly | 70

2. Primary Outcome: Pharmacokinetic Analysis - Total Ribociclib Concentration
Description: Total ribociclib concentrations in non-enhancing and contrast-enhancing tumor tissue samples using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method and equilibrium dialysis
Time Frame: 0-24 hours after the last dose
Measure: Median (Full Range); unit: nanomolar
Groups:
- Ribociclib 400mg Dose: Ribociclib 400mg QD 5 days
- Ribociclib 600mg Dose: Ribociclib 600mg QD 5 days
Arm/Group | Ribociclib 400mg Dose | Ribociclib 600mg Dose
Number analyzed (Participants) | 6 | 18
nanomolar
  Non-Enhancing Tissue | 3132 [1372 to 14954] | 8193 [1314 to 41638]
  Enhancing Tissue | 4056 [2332 to 9900] | 14142 [753 to 49449]

3. Primary Outcome: Pharmacokinetic Analysis - Unbound Ribociclib Concentration
Description: Unbound ribociclib concentrations in non-enhancing and contrast-enhancing tumor tissue samples using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method and equilibrium dialysis
Time Frame: 0-24 hours after the last dose
Measure: Median (Full Range); unit: nanomolar
Arm/Group | Ribociclib 400mg Dose | Ribociclib 600mg Dose
Number analyzed (Participants) | 6 | 18
nanomolar
  Non-Enhancing Tissue | 170 [65 to 1770] | 634 [68 to 2345]
  Enhancing Tissue | 375 [158 to 1405] | 1017 [133 to 4500]

4. Primary Outcome: Pharmacokinetic Analysis - Total Everolimus Concentration
Description: Total everolimus concentrations in non-enhancing and contrast-enhancing tumor tissue samples using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method and equilibrium dialysis
Time Frame: 0-24 hours after the last dose
Measure: Median (Full Range); unit: nanomolar
Groups:
- Everolimus 2.5mg Dose: Everolimus 2.5mg QD 5 days
- Everolimus 5mg Dose: Everolimus 5mg QD 5 days
- Everolimus 10mg Dose: Everolimus 10mg QD 5 days
- Everolimus 50mg Dose: Everolimus 50mg single dose
- Everolimus 60mg Dose: Everolimus 60mg single dose
- Everolimus 70mg Dose: Everolimus 70mg single dose
Arm/Group | Everolimus 2.5mg Dose | Everolimus 5mg Dose | Everolimus 10mg Dose | Everolimus 50mg Dose | Everolimus 60mg Dose | Everolimus 70mg Dose
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3
nanomolar
  Non-Enhancing Tissue | 2.9 [0.2 to 35.3] | 10.3 [9.2 to 20.2] | 4.75 [1.8 to 33.3] | 6.3 [2.4 to 25.1] | 13.8 [11.3 to 36.1] | 8.2 [6.8 to 78.2]
  Enhancing Tissue | 4.4 [0.2 to 83.5] | 16.6 [11.1 to 39.8] | 14.1 [0.2 to 61.3] | 53.05 [1.7 to 74.1] | 30.4 [9.8 to 87.6] | 71.8 [31.2 to 90]

5. Primary Outcome: Pharmacokinetic Analysis - Unbound Everolimus Concentration
Description: Unbound everolimus concentrations in non-enhancing and contrast-enhancing tumor tissue samples using validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method and equilibrium dialysis
Time Frame: 0-24 hours after the last dose
Population: Results are below the lower limit of quantitation (BLQ) (< 0.1 nM)
Measure: Median (Full Range); unit: nanomolar
Arm/Group | Everolimus 2.5mg Dose | Everolimus 5mg Dose | Everolimus 10mg Dose | Everolimus 50mg Dose | Everolimus 60mg Dose | Everolimus 70mg Dose
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3
nanomolar
  Non-Enhancing Tissue | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM)
  Enhancing Tissue | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM) | NA [NA to NA] — Results are below the lower limit of quantitation (BLQ) (< 0.1 nM)

6. Primary Outcome: % Change of pRB+ Cells in Resected Post-Treatment rGMB Tissue vs Baseline Tissue
Description: The percentage change of pRB positive cells in resected post-treatment recurrent GBM tumor tissue compared to baseline (archival primary GBM tumor tissue collected at screening). A positive PD effect is defined as >30% decrease in pRB+ cells.
Time Frame: Baseline, Intraoperatively
Population: 3 participants of 27 enrolled were not included in analysis due to pseudoprogression (dose levels 3, 4, and 6), and an additional 1 participant was excluded due to insufficient tumor content in the resected tissue sample (dose level 6).
Measure: Median (Full Range); unit: Percentage Change of pRB+ Cells
Arm/Group | Dose Level 0: Ribo 400mg+Eve 2.5mg QD | Dose Level 1: Ribo 600mg+Eve 2.5mg QD | Dose Level 2: Ribo 600mg+Eve 5mg QD | Dose Level 3: Ribo 600mg+Eve 10mg QD | Dose Level 4: Ribo 600mg QD+Eve 50mg Once | Dose Level 5: Ribo 600mg QD+Eve 60mg Once | Dose Level 6: Ribo 600mg QD+Eve 70mg Once
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 2
Percentage Change of pRB+ Cells | 34 [-74 to 586] | 25 [-84 to 544] | 268 [24 to 381] | -88 [-98 to -55] | -64 [-90 to 203] | -80 [-85 to 115] | 96 [-74 to 266]

7. Primary Outcome: % Change of pS6+ Cells in Resected Post-Treatment rGMB Tissue vs Baseline Tissue
Description: The percentage change of pS6 positive cells in resected post-treatment recurrent GBM tumor tissue compared to baseline (archival primary GBM tumor tissue collected at screening). A positive PD effect is defined as >30% decrease in pS6+ cells.
Time Frame: Baseline, Intraoperatively
Population: 3 participants of 27 enrolled were not included in analysis due to pseudoprogression (dose levels 3, 4, and 6) and an additional 1 participant was excluded due to insufficient tumor content in the resected tissue sample (dose level 6).
Measure: Median (Full Range); unit: Percentage Change of pS6+ Cells
Arm/Group | Dose Level 0: Ribo 400mg+Eve 2.5mg QD | Dose Level 1: Ribo 600mg+Eve 2.5mg QD | Dose Level 2: Ribo 600mg+Eve 5mg QD | Dose Level 3: Ribo 600mg+Eve 10mg QD | Dose Level 4: Ribo 600mg QD+Eve 50mg Once | Dose Level 5: Ribo 600mg QD+Eve 60mg Once | Dose Level 6: Ribo 600mg QD+Eve 70mg Once
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 3 | 2
Percentage Change of pS6+ Cells | 242 [13 to 423] | -10 [-31 to -4] | 330 [234 to 626] | -8 [-63 to 21] | 431 [-67 to 1365] | -17 [-55 to 88] | -74 [-77 to 88]

8. Secondary Outcome: Median Progression-Free Survival (PFS) in Phase 2 Participants
Description: From date of the first Phase 2 dose until the first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Time Frame: From date of the first Phase 2 dose until the first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Population: No participants were eligible for Phase 2 enrollment
Groups:
- All Phase 2 Participants: All participants who enrolled into the Phase 2 component of the clinical trial.
Arm/Group | All Phase 2 Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Median Overall Survival (OS) in Phase 2 Participants
Description: From date of surgery to date of death from any cause, assessed up to 60 months
Time Frame: From date of surgery to date of death from any cause, assessed up to 60 months
Population: No participants were eligible for Phase 2 enrollment
Arm/Group | All Phase 2 Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Median Concentration of Trough Plasma Concentrations of Total Ribociclib and Total Everolimus in Phase 2 Participants
Description: as for outcome 8
Time Frame: as for outcome 8
Population: No participants were eligible for Phase 2 enrollment
Arm/Group | All Phase 2 Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first date of study drug administration up to 30 days after the last date of study drug administration, assessed up to 37 months
Arm/Group | Dose Level 0: Ribo 400mg+Eve 2.5mg QD | Dose Level 1: Ribo 600mg+Eve 2.5mg QD | Dose Level 2: Ribo 600mg+Eve 5mg QD | Dose Level 3: Ribo 600mg+Eve 10mg QD | Dose Level 4: Ribo 600mg QD+Eve 50mg Once | Dose Level 5: Ribo 600mg QD+Eve 60mg Once | Dose Level 6: Ribo 600mg QD+Eve 70mg Once
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/4 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/3 | 1/3 | 0/4 | 1/4 | 1/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/6 | 3/3 | 1/3 | 3/4 | 2/4 | 2/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: Ribo 400mg+Eve 2.5mg QD (N=6) | Dose Level 1: Ribo 600mg+Eve 2.5mg QD (N=3) | Dose Level 2: Ribo 600mg+Eve 5mg QD (N=3) | Dose Level 3: Ribo 600mg+Eve 10mg QD (N=4) | Dose Level 4: Ribo 600mg QD+Eve 50mg Once (N=4) | Dose Level 5: Ribo 600mg QD+Eve 60mg Once (N=3) | Dose Level 6: Ribo 600mg QD+Eve 70mg Once (N=4)
Brain edema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0: Ribo 400mg+Eve 2.5mg QD (N=6) | Dose Level 1: Ribo 600mg+Eve 2.5mg QD (N=3) | Dose Level 2: Ribo 600mg+Eve 5mg QD (N=3) | Dose Level 3: Ribo 600mg+Eve 10mg QD (N=4) | Dose Level 4: Ribo 600mg QD+Eve 50mg Once (N=4) | Dose Level 5: Ribo 600mg QD+Eve 60mg Once (N=3) | Dose Level 6: Ribo 600mg QD+Eve 70mg Once (N=4)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03834740/Prot_SAP_000.pdf